CLINICAL TRIAL: NCT02594839
Title: A Phase I-II Study to Evaluate Safety and Efficacy of Allogeneic Bone-Marrow Mesenchymal Stem Cells in Patients With Rapidly Progressive Interstitial Lung Disease
Brief Title: Safety and Efficacy of Allogeneic Mesenchymal Stem Cells in Patients With Rapidly Progressive Interstitial Lung Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Federal Research Clinical Center of Federal Medical & Biological Agency, Russia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILD-01
Record Dates: First submitted 2015-11-01; First posted 2015-11-03 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Idiopathic Interstitial Pneumonia; Interstitial Lung Disease; Idiopathic Pulmonary Fibrosis
Keywords: interstitial lung disease; idiopathic interstitial pneumonia; idiopathic pulmonary fibrosis; stem cells
MeSH Terms: conditions — Idiopathic Interstitial Pneumonias; Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MSCs (Experimental): 2 intravenous infusions of suspension of 200 000 000 MSCs each at interval of 7 days. Infusions will be repeated every 3 months for 1 year.
  Interventions: Drug: Bone marrow mesenchymal stem cells
- placebo (Placebo Comparator): 2 intravenous infusions of 400 mL saline each at interval of 7 days. Infusions will be repeated every 3 months for 1 year.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bone marrow mesenchymal stem cells — Bone marrow will be harvested in healthy donors followed by separation and cultivation of MSCs. Before infusion cells will be suspended in 400 mL saline
  Arms: MSCs
Drug: Placebo — intravenous infusion of 400 mL saline
  Arms: placebo

SUMMARY:
The study evaluates the safety and the efficacy of the addition of intravenous transplantation of donor bone marrow mesenchymal stem cells in patients with idiopathic interstitial pneumonia or connective tissue disease associated with interstitial lung disease, which have actively progressing disease with rapid loss of pulmonary function on the background of routine treatment.

DETAILED DESCRIPTION:
Despite significant progress in the treatment of interstitial lung disease, achieved thanks to new drugs, such as pirfenidone and nintedanib, there are many patients for whom these drugs are not available or poorly tolerated. In addition significant evidence of their effectiveness and safety is valid only for idiopathic pulmonary fibrosis. The transplantation of allogeneic stem cells is a promising direction in the modern medicine with the proven safety for different diseases. But the effectiveness of this therapy is still under research. We believe that in most severe cases of a rapidly progressive interstitial lung disease the transplantation of mesenchymal stem cells may be an effective technology due to their immunomodulatory properties.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 20-80 years old
* Diagnosis of idiopathic interstitial pneumonia or secondary to connective tissue diseases interstitial lung disease, based on:

  * Clinical symptoms > 12 months duration,
  * Histologically diagnosed or diagnostic chest HRCT features of interstitial pneumonia
* Forced Vital Capacity (FVC) ≥ 40% predicted and Diffusing Lung Capacity (DLCO) ≥20%
* Loss more than 10% of FVC (L) and DLCO during the last 12 months
* Signed informed consent.

Exclusion Criteria:

* Diagnosis of an interstitial lung disease other than idiopathic interstitial pneumonia or connective tissue disease associated with interstitial lung disease (sarcoidosis, pulmonary alveolar proteinosis, lymphangioleiomyomatosis, pulmonary amyloidosis, exposure-related lung disease etc)
* Obstructive lung disease: FEV1/FVC < 0.70
* Clinically significant medical condition, in the opinion of the investigator, may compromise the results of the study
* Evidence of active infection within 4 week prior to enrollment
* History of malignancy < 5 years prior to enrollment
* Unable to cooperate with any study procedures
* Pregnant or breast-feeding
* Treatment with antiinflammatory or antifibrotic drugs including oral steroids, cytostatic drugs, pirfenidone, D penicillamine, colchicine, tumor necrosis factor α blockers, imatinib, interferon γ, monoclonal antibodies < 6 months prior to randomization.
* Active listing for transplant of any organ.
* Known history of alcohol abuse within 1 year prior to enrollment
* Participation in another clinical trial

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Safety: Number of serious adverse events | 12 months
  registration of adverse events related to infusion and 12 months follow-up

SECONDARY OUTCOMES:
DLCO changes from baseline | 12 months
  Assessment of the diffusing lung capacity at 3, 6, 9, 12 months of treatment
FVC changes from baseline | 12 months
  Assessment of spirometry at 3, 6, 9, 12 months of treatment
exercise capacity changes | 12 months
  Assessment of 6MWD at 3, 6, 9, 12 months of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Federal Research Clinical Center FMBA of Russia, Moscow, Russia